CLINICAL TRIAL: NCT03346434
Title: A Phase 2/3 Study Investigating the Pharmacokinetics, Safety, and Efficacy of Dupilumab in Patients Aged ≥6 Months to <6 Years With Moderate-to-Severe Atopic Dermatitis
Brief Title: Safety, Pharmacokinetics and Efficacy of Dupilumab in Patients ≥6 Months to <6 Years With Moderate-to-Severe Atopic Dermatitis (Liberty AD PRESCHOOL)
Acronym: Liberty AD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R668-AD-1539; 2016-000955-28 (EudraCT Number)
Record Dates: First submitted 2017-02-06; First posted 2017-11-17 (Actual); Results first posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Dermatitis, Atopic
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: Part A: Single-ascending-dose cohorts staggered by age;
  Part B: Parallel Group
Masking Description: Part A: Open Label;
  Part B: Masked, Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A (Open label Dupilumab): Age cohorts 1 & 2 (Experimental): Age cohort 1: ≥2 years old to <6 years old
  Age cohort 2: ≥6 months to <2 years old
  Interventions: Drug: Dupilumab
- Part B (Double-blind): Dupilumab dose 1 (Experimental): The results of part A will be used to guide the selection of dose levels and dosing frequency for part B.
  Interventions: Drug: Dupilumab
- Part B (Double-blind): Dupilumab dose 2 (Experimental): The results of part A will be used to guide the selection of dose levels and dosing frequency for part B.
  Interventions: Drug: Dupilumab
- Part B (Double-Blind): Placebo (Experimental)
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Dupilumab — Solution for injection, subcutaneous (SC)
  Other Names: DUPIXENT®; REGN668; SAR231893
  Arms: Part A (Open label Dupilumab): Age cohorts 1 & 2; Part B (Double-blind): Dupilumab dose 1; Part B (Double-blind): Dupilumab dose 2
Drug: Matching placebo — Solution for injection, subcutaneous (SC)
  Arms: Part B (Double-Blind): Placebo

SUMMARY:
This study is a 2-part (parts A and B) phase 2/3 study to evaluate the safety, pharmacokinetics (PK) and efficacy of dupilumab in participants 6 months to less than 6 years of age with moderate-to-severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
1. Part A (open-label, single-ascending-dose, sequential cohort phase 2 study):

   * Primary objective is to characterize the safety and PK of dupilumab administered as a single dose in pediatric participants, 6 months to less than 6 years of age, with severe AD.
   * Secondary objective is to evaluate the efficacy and immunogenicity of a single dose of dupilumab in participants 6 months to less than 6 years of age with severe AD.
2. Part B (randomized, double-blind, parallel-group, placebo-controlled phase 3 study):

   * Primary objective is to demonstrate the efficacy of multiple doses of dupilumab over 16 weeks of treatment when administered concomitantly with topical corticosteroids (TCS) in pediatric participants, 6 months to less than 6 years of age, with moderate-to-severe AD.
   * Secondary objective is to assess the safety and immunogenicity of multiple doses of dupilumab over 16 weeks of treatment when administered concomitantly with TCS in participants 6 months to less than 6 years of age with moderate-to-severe AD.

ELIGIBILITY:
Key Inclusion Criteria

* Diagnosis of atopic dermatitis (AD) according to the American Academy of Dermatology consensus criteria at the screening visit
* Participants with documented recent history (within 6 months before the screening visit) of inadequate response to topical AD medication(s)
* IGA score at screening and baseline visits
* part A: IGA = 4
* part B: IGA ≥3
* EASI score at screening and baseline visits
* part A: EASI ≥21
* part B: EASI ≥16
* Body Surface Area (BSA) involvement at screening and baseline visits
* part A: ≥15%
* part B: ≥10%
* At least 11 (of a total of 14*) applications of a topical emollient (moisturizer) during the 7 consecutive days immediately before the baseline visit (not including the day of randomization) (for part B of the study only)
* Baseline worst scratch/itch score weekly average score for maximum scratch/itch intensity ≥4 (for part B of the study only)
* At least 11 (of a total of 14) daily applications of low potency TCS during the 2-week TCS standardization period (beginning on day -14) leading up to the baseline visit (for part B of the study only).

Key Exclusion Criteria

* Prior treatment with dupilumab
* History of important side effects of low potency topical corticosteroids (only applicable for part B of the study)
* Having used immunosuppressive/immunomodulating drugs within 4 weeks before the baseline visit
* Treatment with a live (attenuated) vaccine within 4 weeks before the baseline visit
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiprotozoals, or antifungals within 2 weeks before the baseline visit.
* Known or suspected immunodeficiency, known history of human immunodeficiency virus (HIV) infection or HIV seropositivity at the screening visit, established diagnosis of HBV infection or HBV seropositivity at screening, established diagnosis of HCV infection or HCV seropositivity at screening
* History of malignancy at any time before the baseline visit
* Diagnosed active endoparasitic infections or at high risk of these infections
* Severe concomitant illness(es) that, in the investigator's judgment, would adversely affect the patient's participation in the study
* Body weight <5 kg or ≥30 kg at baseline (only applicable part B of the study)

Note: Other protocol defined Inclusion/ Exclusion criteria apply

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 202 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (47):
- United States (33):
  - Regeneron Investigational Site, Birmingham, Alabama
  - Regeneron Investigational Site, Gilbert, Arizona
  - Regeneron Investigational Site, Long Beach, California
  - Regeneron Investigational site, Los Angeles, California
  - Regeneron Investigational Site, Palo Alto, California
  - Regeneron Investigational Site, Rolling Hills Estates, California
  - Regeneron Investigational Site, San Diego, California
  - Regeneron Investigational Site, Washington D.C., District of Columbia
  - Regeneron Investigational Site, Coral Gables, Florida
  - Regeneron Investigational Site, Tampa, Florida
  - Regeneron Investigational Site, Columbus, Georgia
  - Regeneron Investigational Site, Macon, Georgia
  - Regeneron Investigational Site, Sandy Springs, Georgia
  - Regeneron Investigational Site, Chicago, Illinois
  - Regeneron Investigational Site, Rockville, Maryland
  - Regeneron Investigational Site, Boston, Massachusetts
  - Regeneron Investigational Site, Ann Arbor, Michigan
  - Regeneron Investigational Site, Ypsilanti, Michigan
  - Regeneron Investigational Site, St Louis, Missouri
  - Regeneron Investigational Site, Lincoln, Nebraska
  - Regeneron Investigational Site, Hackensack, New Jersey
  - Regeneron Investigational Site, Forest Hills, New York
  - Regeneron Investigational Site, New York, New York
  - Regeneron Investigational Site, Rochester, New York
  - Regeneron Investigational Site, Portland, Oregon
  - Regeneron Investigational Site, Philadelphia, Pennsylvania
  - Regeneron Investigational Site, Charleston, South Carolina
  - Regeneron Investigational Site, North Charleston, South Carolina
  - Regeneron Investigational Site, Austin, Texas
  - Regeneron Investigational Site, San Antonio, Texas
  - Regeneron Investigational Site, Norfolk, Virginia
  - Regeneron Investigational Site, Seattle, Washington
  - Regeneron Investigational Site, Milwaukee, Wisconsin
- Germany (7):
  - Regeneron Investigational Site, Osnabrück, Lower Saxony
  - Regeneron Investigational site, Münster, North Rhine-Westphal
  - Regeneron Investigational Site, Dresden, Saxony
  - Regeneron Investigational site, Frankfurt am Main
  - Regeneron Investigational Site, Kiel
  - Regeneron Investigational Site, München
  - Regeneron Investigational site, München
- Poland (5):
  - Regeneron Investigational Site, Bialystok
  - Regeneron Investigational Site, Katowice
  - Regeneron Investigational Site, Krakow
  - Regeneron Investigational Site, Ostrowiec Świętokrzyski
  - Regeneron Investigational Site, Warsaw
- United Kingdom (2):
  - Regeneron Investigational Site, Manchester, Lancashire
  - Regeneron Investigational Site, Sheffield, South Yorkshire

REFERENCES:
- [Derived] Langley RG, Gherardi G, Coleman A, Ardeleanu M, Rodriguez-Marco A, Levy S, Bansal A, Chen Z, Rossi AB, Shumel B, Khokhar FA. The Safety Data of Dupilumab for the Treatment of Moderate-to-Severe Atopic Dermatitis in Infants, Children, Adolescents, and Adults. Am J Clin Dermatol. 2025 Nov;26(6):981-1002. doi: 10.1007/s40257-025-00952-w. Epub 2025 Sep 24. PMID 40993471
- [Derived] Rossi AB, Mello AM, Zahn J. Dupilumab Efficacy in Children with Atopic Dermatitis with Different Phenotypes and Endotypes: A Case Series. Adv Ther. 2025 Jul;42(7):3186-3206. doi: 10.1007/s12325-025-03150-6. Epub 2025 May 8. PMID 40338484
- [Derived] Kamal MA, Kosloski MP, Lai CH, Partridge MA, Rajadhyaksha M, Kanamaluru V, Bansal A, Shabbir A, Shumel B, Ardeleanu M, Richards SM, Yan H, Xu CR, Rodriguez-Marco A, Xiao J, Khokhar FA, Gherardi G, Babilonia E, Maloney J, Mortensen E, Akinlade B, Braunstein N, Stahl N, Torri A, Davis JD, DiCioccio AT. Immunogenicity of dupilumab in adult and pediatric patients with atopic dermatitis. Front Immunol. 2024 Nov 11;15:1466372. doi: 10.3389/fimmu.2024.1466372. eCollection 2024. PMID 39588375
- [Derived] Boguniewicz M, Sher LD, Paller AS, Arkwright PD, Yoshihara S, Chen Z, Shah P, Marco AR. Dupilumab is Efficacious in Young Children with Atopic Dermatitis Regardless of Type 2 Comorbidities. Adv Ther. 2024 Dec;41(12):4601-4616. doi: 10.1007/s12325-024-02998-4. Epub 2024 Oct 29. PMID 39470878
- [Derived] Paller AS, Siegfried EC, Simpson EL, Cork MJ, Sidbury R, Chen IH, Khokhar FA, Xiao J, Dubost-Brama A, Bansal A. Dupilumab Safety and Efficacy up to 1 Year in Children Aged 6 Months to 5 Years with Atopic Dermatitis: Results from a Phase 3 Open-Label Extension Study. Am J Clin Dermatol. 2024 Jul;25(4):655-668. doi: 10.1007/s40257-024-00859-y. Epub 2024 May 14. PMID 38743155
- [Derived] Paller AS, Siegfried EC, Cork MJ, Arkwright PD, Eichenfield LF, Ramien M, Khokhar FA, Chen Z, Zhang A, Cyr SL. Infections in Children Aged 6 Months to 5 Years Treated with Dupilumab in a Placebo-Controlled Clinical Trial of Moderate-to-Severe Atopic Dermatitis. Paediatr Drugs. 2024 Mar;26(2):163-173. doi: 10.1007/s40272-023-00611-9. Epub 2024 Jan 24. PMID 38267692
- [Derived] Paller AS, Pinter A, Wine Lee L, Aschoff R, Zdybski J, Schnopp C, Praestgaard A, Bansal A, Shumel B, Prescilla R, Bastian M. Efficacy and Safety of Dupilumab Treatment with Concomitant Topical Corticosteroids in Children Aged 6 Months to 5 Years with Severe Atopic Dermatitis. Adv Ther. 2024 Mar;41(3):1046-1061. doi: 10.1007/s12325-023-02753-1. Epub 2024 Jan 9. PMID 38194047
- [Derived] Siegfried EC, Simpson EL, Cork MJ, Arkwright PD, Wine Lee L, Chen Z, Prescilla R, Bansal A, Levit NA, Rodriguez Marco A. Dupilumab Treatment Leads to Rapid and Consistent Improvement of Atopic Dermatitis in All Anatomical Regions in Patients Aged 6 Months to 5 Years. Dermatol Ther (Heidelb). 2023 Sep;13(9):1987-2000. doi: 10.1007/s13555-023-00960-w. Epub 2023 Jul 22. PMID 37480432
- [Derived] Yang N, Ye Y, Shao J, Wu H, Xu Q, Zhu J, Liu J, Li Z. Efficacy of Dupilumab in Children 6 Months to 11 Years Old With Atopic Dermatitis: A Retrospective Real-World Study in China. Dermatitis. 2024 Jan-Feb;35(S1):S39-S46. doi: 10.1089/derm.2022.0069. Epub 2023 Feb 17. PMID 36800177
- [Derived] Paller AS, Siegfried EC, Cork MJ, Wollenberg A, Arkwright PD, Gonzalez ME, Lockshin B, Chen Z, Bansal A, Levit NA, Prescilla R. Laboratory Safety from a Randomized 16-Week Phase III Study of Dupilumab in Children Aged 6 Months to 5 Years with Moderate-to-Severe Atopic Dermatitis. Paediatr Drugs. 2023 Jan;25(1):67-77. doi: 10.1007/s40272-022-00553-8. Epub 2022 Dec 19. PMID 36529811
- [Derived] Paller AS, Simpson EL, Siegfried EC, Cork MJ, Wollenberg A, Arkwright PD, Soong W, Gonzalez ME, Schneider LC, Sidbury R, Lockshin B, Meltzer S, Wang Z, Mannent LP, Amin N, Sun Y, Laws E, Akinlade B, Dillon M, Kosloski MP, Kamal MA, Dubost-Brama A, Patel N, Weinreich DM, Yancopoulos GD, O'Malley JT, Bansal A; participating investigators. Dupilumab in children aged 6 months to younger than 6 years with uncontrolled atopic dermatitis: a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2022 Sep 17;400(10356):908-919. doi: 10.1016/S0140-6736(22)01539-2. PMID 36116481

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 2 parts: Part A and Part B; Participants who enrolled in Part A of study were not eligible to participate in Part B.
Pre-assignment Details: Participants in Part A enrolled in 2 sequential age cohorts: Cohort 1 (≥2 to <6 yrs) and Cohort 2 (≥6 months to <2 yrs). Each age cohort received dupilumab in 1 of 2 doses: 3 milligrams per kilogram (mg/kg) or 6 mg/kg. Participants in Part B were randomized to 1 of 2 treatment groups: placebo + topical corticosteroids (TCS) or dupilumab 200/300 mg every four weeks (Q4W) + TCS.
Groups:
- Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg: Participants received a single subcutaneous (SC) injection of dupilumab at a dose of 3 mg/kg at Day 1. At week 4, participants could roll over into an open-label extension (OLE) study (R668-AD-1434/NCT02612454), if considered eligible. Participants who did not enter the OLE study were followed for up to an additional 4 weeks for safety.
- Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg; Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg: Participants received a single SC injection of dupilumab at a dose of 6 mg/kg at Day 1. At week 4, participants could roll over into an OLE study (R668-AD-1434/NCT02612454), if considered eligible. Participants who did not enter the OLE study were followed for up to an additional 4 weeks for safety.
- Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg: Participants received a single SC injection of dupilumab at a dose of 3 mg/kg at Day 1. At week 4, participants could roll over into an OLE study (R668-AD-1434/NCT02612454), if considered eligible. Participants who did not enter the OLE study were followed for up to an additional 4 weeks for safety.
- Part B: Placebo + TCS: Participants received SC injection of placebo matched to dupilumab Q4W for 16 weeks along with low potency TCS applied once daily to areas with active lesions. At week 16, participants could roll over into an OLE study (R668-AD-1434/ NCT02612454), if considered eligible. Participants who did not enter the OLE study were followed for up to an additional 12 weeks for safety (Week 28, end of study [EOS] period).
- Part B: Dupilumab 200 mg or 300 mg Q4W + TCS: Participants with baseline weight of ≥ 5 to < 15 kilogram (kg) received SC injections of 200 mg or participants with baseline weight ≥ 15 to < 30 kg received SC injections of 300 mg of dupilumab at Day 1 and Q4W from week 4 to week 12. Participants applied low potency TCS once daily to areas with active lesions for 16 weeks. At week 16, participants could roll over into an OLE study (R668-AD-1434/NCT02612454), if considered eligible. Participants who did not enter the OLE study were followed for up to an additional 12 weeks for safety (Week 28, EOS period).
Period: Overall Study
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Started | 10 | 10 | 10 | 10 | 79 | 83
Completed Part A | 10 | 10 | 9 | 10 | 0 | 0
Completed Part B (Week 16) | 0 | 0 | 0 | 0 | 76 | 83
Completed Part B (Week 28) (End of Study) | 0 | 0 | 0 | 0 | 1 | 1
Completed | 10 | 10 | 9 | 10 | 1 | 1
Not Completed | 0 | 0 | 1 | 0 | 78 | 82
Not completed — Randomized in Error | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Transitioned to OLE study at Week 16 (NCT02612454) | 0 | 0 | 0 | 0 | 75 | 81

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 79 | 83 | 202
Age, Customized [Number; unit: Participants]
  6 months - <2 years | 0 | 0 | 10 | 10 | 5 | 6 | 31
  ≥2 years and <6 years | 10 | 10 | 0 | 0 | 74 | 77 | 171
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 2 | 24 | 39 | 73
  Male | 6 | 7 | 9 | 8 | 55 | 44 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 2 | 9 | 11 | 29
  Not Hispanic or Latino | 7 | 8 | 8 | 8 | 70 | 72 | 173
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigator Global Assessment (IGA) [Count of Participants; unit: Participants] — The IGA is an assessment scale used in clinical studies to rate the severity of atopic dermatitis (AD) globally, based on a 5-point scale ranging from 0 to 4 where 0=clear; 1=almost clear; 2=mild; 3=moderate; 4=severe.
  Participants
    IGA=3 (moderate) | 0 | 0 | 0 | 0 | 17 | 20 | 37
    IGA=4 (severe) | 10 | 10 | 10 | 10 | 62 | 63 | 165

OUTCOME MEASURES:

1. Primary Outcome: Part A: Maximum Observed Serum Concentration (Cmax) of Functional Dupilumab
Description: Serum concentration of functional dupilumab was reported.
Time Frame: Post-dose on Days 1, 3, 8, 18, and 29
Population: The Pharmacokinetic Analysis Set (PKAS) included all treated participants who received any study drug (safety analysis set) and who had at least 1 non-missing functional dupilumab measurement following the administration of the first dose of study drug.
Measure: Mean (Standard Deviation); unit: Milligrams per Liter (mg/L)
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg
Number analyzed (Participants) | 9 | 10 | 10 | 10
Milligrams per Liter (mg/L) | 25.2 (7.44) [lower limit 7.44] | 49.8 (11.3) [lower limit 11.3] | 20.1 (6.81) [lower limit 6.81] | 46.1 (11.1) [lower limit 11.1]

2. Primary Outcome: Part A: Dose Normalized Maximum Observed Serum Concentration (Cmax/Dose) of Dupilumab
Description: Dose normalized was calculated as Cmax obtained directly from the concentration versus time curve divided by dose. Cmax/dose was measured in Milligrams per Liter/Milligrams per Kilogram ([mg/L]/[mg/kg]).
Time Frame: Post-dose on Days 1, 3, 8, 18, and 29
Population: The PKAS included all treated participants who received any study drug (safety analysis set) and who had at least 1 non-missing functional dupilumab measurement following the administration of the first dose of study drug.
Measure: Mean (Standard Deviation); unit: [mg/L]/[mg/kg]
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg
Number analyzed (Participants) | 9 | 10 | 10 | 10
[mg/L]/[mg/kg] | 8.39 (2.48) [lower limit 2.48] | 8.30 (1.89) [lower limit 1.89] | 6.70 (2.27) [lower limit 2.27] | 7.68 (1.86) [lower limit 1.86]

3. Primary Outcome: Part A: Time to Reach the Maximum Serum Concentration (Tmax) of Dupilumab
Description: Tmax was obtained directly from the concentration versus time curve.
Time Frame: Post-dose on Days 1, 3, 8, 18, and 29
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg
Number analyzed (Participants) | 10 | 10 | 10 | 9
Days | 1.97 (1.87) [1.87 to 7.82] | 1.95 (1.75) [1.75 to 3.08] | 2.10 (1.80) [1.80 to 7.99] | 1.92 (1.72) [1.72 to 3.02]

4. Primary Outcome: Part A: Last Quantifiable Serum Concentration (Clast) of Dupilumab
Description: Clast is the last measurable serum concentration of dupilumab.
Time Frame: Post-dose on Days 1, 3, 8, 18, and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg
Number analyzed (Participants) | 9 | 10 | 10 | 10
mg/L | 6.64 (6.16) [lower limit 6.16] | 6.14 (4.69) [lower limit 4.69] | 5.64 (4.52) [lower limit 4.52] | 15.1 (9.48) [lower limit 9.48]

5. Primary Outcome: Part A: Time of the Last Quantifiable Serum Concentration (Tlast) of Dupilumab
Description: Tlast was defined as the last time point with a measurable serum concentration of dupilumab.
Time Frame: Post-dose on Days 1, 3, 8, 18, and 29
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg
Number analyzed (Participants) | 9 | 10 | 10 | 10
Days | 14.8 (6.79) [6.79 to 28.0] | 26.5 (15.0) [15.0 to 32.0] | 8.56 (6.88) [6.88 to 16.9] | 16.0 (6.95) [6.95 to 28.0]

6. Primary Outcome: Part A: Area Under the Serum Concentration-Time Curve From Time Zero to the Time of the Last Measurable Concentration (AUClast) of Dupilumab
Description: AUClast was defined as area under the serum concentration time-curve from zero to the last measured concentration.
Time Frame: Post-dose on Days 1, 3, 8, 18, and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days*Milligrams per Liter (day*mg/L)
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg
Number analyzed (Participants) | 9 | 10 | 10 | 10
Days*Milligrams per Liter (day*mg/L) | 198 (125) [lower limit 125] | 622 (184) [lower limit 184] | 123 (86.0) [lower limit 86.0] | 493 (294) [lower limit 294]

7. Primary Outcome: Part A: Dose Normalized Area Under the Serum Concentration-Time Curve From Time Zero to the Time of the Last Measurable Concentration (AUClast/Dose) of Dupilumab
Description: Dose normalized AUClast was calculated by AUClast/dose.
Time Frame: Post-dose on Days 1, 3, 8, 18, and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: [day*mg/L]/[mg/kg]
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg
Number analyzed (Participants) | 9 | 10 | 10 | 10
[day*mg/L]/[mg/kg] | 66.0 (41.6) [lower limit 41.6] | 104 (30.6) [lower limit 30.6] | 41.0 (28.7) [lower limit 28.7] | 82.1 (48.9) [lower limit 48.9]

8. Primary Outcome: Part A: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: Adverse Event (AE) was defined as any untoward medical occurrence in a participant administered a study drug which may/may not have a causal relationship with study drug. Serious AE (SAE) was defined as any untoward medical occurrence that resulted in any of following outcomes: death, life-threatening, required initial/prolonged in-participant hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect/considered as medically important event. TEAE was defined as AE starting/worsening after first intake of study drug. TEAEs included participants with both SAEs and non-SAEs. Number of participants with TEAEs is reported.
Time Frame: Baseline up to Week 4
Population: The safety analysis set (SAF) included all participants who received any study drug and were analyzed based on the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg
Number analyzed (Participants) | 10 | 10 | 10 | 10
Participants | 3 | 2 | 7 | 7

9. Primary Outcome: Part A: Number of Participants With TEAEs by Severity According to Qualitative Toxicity Scale
Description: Severity of TEAEs were graded using Qualitative Toxicity Scale, as follows: Mild: Participant is aware of the event or symptom, but the event or symptom is easily tolerated; Moderate: Participant experiences sufficient discomfort to interfere with or reduce his or her usual level of activity; Severe: Significant impairment of functioning: the participant is unable to carry out his or her usual activities. Number of participants with TEAEs by severity were reported.
Time Frame: Baseline up to Week 4
Population: The SAF included all participants who received any study drug and were analyzed based on the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg
Number analyzed (Participants) | 10 | 10 | 10 | 10
Participants
  Mild | 1 | 2 | 4 | 5
  Moderate | 2 | 0 | 2 | 2
  Severe | 0 | 0 | 1 | 0

10. Primary Outcome: Part B: Percentage of Participants With Investigator's Global Assessment (IGA) Score 0 or 1 at Week 16
Description: The IGA is an assessment scale used in clinical studies to rate the severity of AD globally, based on a 5-point scale ranging from 0 to 4 where 0 = clear; 1=almost clear; 2=mild; 3=moderate; 4=severe. A negative change from baseline indicated improvement. Percentage of participants with IGA score of '0' or '1' is reported.
Time Frame: Week 16
Population: The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized). Missing data due to withdrawn consent, adverse event (AE), lack of efficacy were imputed as non responder. Missing data due to any other reason including COVID-19 were imputed using multiple imputation (MI). Participants were considered as non-responders after initiation of rescue treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 79 | 83
Percentage of Participants | 3.9 (-0.42) [-0.42 to 8.21] | 27.7 (18.45) [18.45 to 38.62]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 23.8, 95% CI 2-sided [13.27 to 34.37]

11. Primary Outcome: Part B: Percentage of Participants With Eczema Area and Severity Index (EASI) -75 (EASI-75) (≥75% Improvement From Baseline) at Week 16
Description: The EASI score is used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper, and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores indicating the worse severity of AD. EASI-75 responders were the participants who achieved ≥75% overall improvement in EASI score from baseline at Week 16.
Time Frame: Week 16
Population: The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized). Missing data due to withdrawn consent, AE, lack of efficacy were imputed as non responder. Missing data due to any other reason including COVID-19 were imputed using MI. Participants were considered as non-responders after initiation of rescue treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 79 | 83
Percentage of Participants | 10.7 (3.65) [3.65 to 17.74] | 53.0 (41.74) [41.74 to 64.07]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 42.3, 95% CI 2-sided [29.47 to 55.16]

12. Secondary Outcome: Part A: Number of Participants With Serious TEAEs and Severe TEAEs
Description: Adverse Event (AE) was defined as any untoward medical occurrence in a participant administered a study drug which may/may not have a causal relationship with study drug. A serious TEAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. Severe TEAE: significant impairment of functioning the participant is unable to carry out his or her usual activities.
Time Frame: Baseline up to Week 4
Population: The SAF included all participants who received any study drug and was analyzed based on the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg
Number analyzed (Participants) | 10 | 10 | 10 | 10
Participants
  Participants with serious TEAEs | 1 | 0 | 1 | 0
  Participants with severe TEAEs | 0 | 0 | 1 | 0

13. Secondary Outcome: Part A: Percent Change From Baseline in EASI Score at Week 4
Description: The EASI score is used to measure the severity and extent of AD and measured erythema, infiltration, excoriation, and lichenification on 4 anatomic regions of the body: head, trunk, upper, and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores indicated the worse severity of AD. A negative change from baseline indicated improvement.
Time Frame: Week 4
Population: The SAF included all participants who received any study drug and was analyzed based on the actual treatment received.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg
Number analyzed (Participants) | 10 | 10 | 10 | 10
Percent Change | -26.6 (47.37) [lower limit 47.37] | -48.7 (28.89) [lower limit 28.89] | -22.4 (42.52) [lower limit 42.52] | -43.2 (35.55) [lower limit 35.55]

14. Secondary Outcome: Part A: Percent Change From Baseline in SCORing Atopic Dermatitis (SCORAD) Score at Week 4
Description: The SCORAD is used to assess the extent and severity of AD. Extent and severity of eczema as well as subjective symptoms (insomnia, etc) were assessed and scored. SCORAD total score ranges from 0 (absent disease) to 103 (severe disease). A negative change from baseline indicated improvement.
Time Frame: Week 4
Population: SAF included all participants who received any study drug and was analyzed based on the actual treatment received.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg
Number analyzed (Participants) | 10 | 10 | 10 | 10
Percent Change | -18.6 (26.18) [lower limit 26.18] | -31.9 (17.45) [lower limit 17.45] | -22.4 (26.44) [lower limit 26.44] | -28.1 (27.84) [lower limit 27.84]

15. Secondary Outcome: Part A: Percentage of Participants With IGA Score 0 or 1 at Week 4
Description: The IGA is an assessment scale used in clinical studies to rate the severity of AD globally, based on a 5-point scale ranging from 0 to 4 where 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe. Percentage of participants with IGA score of '0' or '1' were reported.
Time Frame: Week 4
Population: SAF included all participants who received any study drug and was analyzed based on the actual treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg
Number analyzed (Participants) | 10 | 10 | 10 | 10
Percentage of Participants | 10.0 (0.25) [0.25 to 44.50] | 0.0 (0.00) [0.00 to 30.85] | 10.0 (0.25) [0.25 to 44.50] | 10.0 (0.25) [0.25 to 44.50]

16. Secondary Outcome: Part A: Number of Participants With at Least One Positive Treatment-Emergent Anti-Drug Antibodies (ADA)
Description: Treatment boosted (TB) Response: Any post-dose positive result at least 9-fold over the baseline level when baseline is positive; Treatment emergent (TE) Response: Post-dose positive result when baseline results were negative.
Time Frame: Baseline up to Day 57
Population: The ADA Analysis Set (AAS) included all treated participants who received any study drug and who had at least 1 non-missing ADA result following the first dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg
Number analyzed (Participants) | 10 | 10 | 10 | 10
Participants
  TB Response | 0 | 0 | 1 | 0
  TE Response | 5 | 4 | 5 | 5

17. Secondary Outcome: Part B: Number of Participants With at Least One Serious Adverse Event (SAE) Through Week 16
Time Frame: Baseline through Week 16
Population: SAF included all randomized participants who received at least one dose of study drug and was analysed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 78 | 83
Participants | 4 | 0

18. Secondary Outcome: Part B: Number of Participants With at Least One Skin Infection Treatment Emergent Adverse Event (TEAE) (Excluding Herpetic Infection) Through Week 16
Time Frame: Baseline through Week 16
Population: SAF included all randomized participants who received at least one dose of study drug and was analysed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 78 | 83
Participants | 19 | 10

19. Secondary Outcome: Part B: Number of Participants With at Least One Positive Treatment-Emergent ADA
Description: Treatment emergent (TE): Post-dose positive result when baseline results were negative.
Time Frame: Baseline up to Day 197
Population: AAS included all participants who received any study drug and who had at least one non-missing ADA result after the first dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 69 | 74
Participants | 0 | 1

20. Secondary Outcome: Part B: Percent Change From Baseline in EASI Score at Week 16
Description: The EASI score is used to measure the severity and extent of AD and measures erythema, infiltration, excoriation, and lichenification on 4 anatomic regions of the body: head, trunk, upper, and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores indicating the worse severity of AD. A negative change from baseline indicated improvement.
Time Frame: Week 16
Population: FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomisation (as randomised). Missing data due to withdrawn consent, AE, or lack of efficacy and data after rescue were imputed by post baseline worst observation carried forward (WOCF). If there was no post baseline assessment, the baseline value was used. Missing values due to other reasons including COVID-19 were imputed by MI approach.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 79 | 83
Percent Change | -19.6 (5.13) [lower limit 5.13] | -70.0 (4.85) [lower limit 4.85]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; Least Square (LS) Mean Difference = -50.4, 95% CI 2-sided [-62.38 to -38.40]

21. Secondary Outcome: Part B: Percent Change From Baseline in Weekly Average of Daily Worst Scratch/Itch/Numerical Rating Scale (NRS) at Week 16
Description: Pruritus NRS is an assessment tool used to report intensity of participant's pruritus (itch), both average & maximum intensity, during 24-hr recall period. Participants were asked two questions: 1) For average itch intensity: how would you rate your itch overall (on average) during the previous 24 hrs; 2) For maximum itch intensity: How would you rate your itch at the worst moment during the previous 24 hrs? Both questions were rated on a scale: 0-10 with 0=no itch & 10=worst itch imaginable. A negative change from baseline indicated improvement.
Time Frame: Week 16
Population: The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized). Missing data due to withdrawn consent, AE, or lack of efficacy and data after rescue were imputed by post baseline WOCF. If there was no post baseline assessment, the baseline value was used. Missing values due to other reasons including COVID-19 were imputed by MI approach.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 79 | 83
Percent Change | -2.2 (5.22) [lower limit 5.22] | -49.4 (5.03) [lower limit 5.03]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -47.1, 95% CI 2-sided [-59.47 to -34.79]

22. Secondary Outcome: Part B: Percentage of Participants With Improvement (Reduction From Baseline) of Weekly Average of Daily Worst Scratch/Itch/NRS ≥4 Points at Week 16
Description: Pruritus NRS is an assessment tool used to report intensity of subject's pruritus (itch), both average & maximum intensity, during 24-hr recall period. Subjects were asked two questions: 1) For average itch intensity: how would you rate your itch overall (on average) during the previous 24 hrs; & 2) For maximum itch intensity: How would you rate your itch at the worst moment during the previous 24 hrs? Both questions were rated on a scale: 0-10 with 0=no itch & 10=worst itch imaginable.
Time Frame: Week 16
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 78 | 83
Percentage of Participants | 8.9 (2.25) [2.25 to 15.51] | 48.1 (37.05) [37.05 to 59.15]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 39.2, 95% CI 2-sided [26.18 to 52.27]

23. Secondary Outcome: Part B: Percentage of Participants With Improvement (Reduction From Baseline) of Weekly Average of Daily Worst Scratch/Itch/NRS ≥3 Points at Week 16
Description: Pruritus NRS is an assessment tool used to report intensity of participant's pruritus (itch), both average & maximum intensity, during 24-hr recall period. Participants were asked two questions: 1) For average itch intensity: how would you rate your itch overall (on average) during the previous 24 hrs; & 2) For maximum itch intensity: How would you rate your itch at the worst moment during the previous 24 hrs? Both questions were rated on a scale: 0-10 with 0=no itch & 10=worst itch imaginable.
Time Frame: Week 16
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 78 | 83
Percentage of Participants | 9.9 (2.59) [2.59 to 17.22] | 53.3 (42.29) [42.29 to 64.22]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 43.3, 95% CI 2-sided [30.03 to 56.67]

24. Secondary Outcome: Part B: Percentage of Participants Who Achieved EASI-50 (≥50% Improvement From Baseline) at Week 16
Description: The EASI score is used to measure the severity and extent of AD and measured erythema, infiltration, excoriation, and lichenification on 4 anatomic regions of the body: head, trunk, upper, and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores indicating the worse severity of AD. EASI-50 responders were the participants who achieved ≥50% overall improvement in EASI score from baseline at Week 16.
Time Frame: Week 16
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 79 | 83
Percentage of Participants | 20.2 (11.09) [11.09 to 29.23] | 68.7 (57.56) [57.56 to 78.41]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 48.5, 95% CI 2-sided [35.03 to 62.00]

25. Secondary Outcome: Part B: Percentage of Participants Who Achieved EASI-90 (≥90% Improvement From Baseline) at Week 16
Description: The EASI score is used to measure the severity and extent of AD and measured erythema, infiltration, excoriation, and lichenification on 4 anatomic regions of the body: head, trunk, upper, and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores indicating the worse severity of AD. EASI-90 responders were the participant who achieved ≥90% overall improvement in EASI score from baseline at Week 16.
Time Frame: Week 16
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 79 | 83
Percentage of Participants | 2.8 (-1.02) [-1.02 to 6.66] | 25.3 (16.39) [16.39 to 36.04]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 22.5, 95% CI 2-sided [12.37 to 32.60]

26. Secondary Outcome: Part B: Change From Baseline in Percent Body Surface Area (BSA) Affected by Atopic Dermatitis (AD) at Week 16
Description: BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined. A negative change from baseline indicated improvement.
Time Frame: Week 16
Population: The FAS included all randomized participant. Efficacy analyses were based on the treatment allocated at randomization (as randomized). Missing data due to withdrawn consent, AE, or lack of efficacy and data after rescue were imputed by post baseline WOCF. If there was no post baseline assessment, the baseline value was used. Missing values due to other reasons including COVID-19 were imputed by MI approach.
Measure: Least Squares Mean (Standard Error); unit: Percentage of Body Surface Area (BSA)
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 79 | 83
Percentage of Body Surface Area (BSA) | -10.74 (2.926) [lower limit 2.926] | -35.00 (2.815) [lower limit 2.815]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -24.27, 95% CI 2-sided [-31.204 to -17.329]

27. Secondary Outcome: Part B: Change From Baseline in Patient Oriented Eczema Measure (POEM) at Week 16
Description: The POEM is a 7-item questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]). A negative change from baseline indicated improvement.
Time Frame: Week 16
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 79 | 83
Score on a Scale | -3.8 (0.92) [lower limit 0.92] | -12.9 (0.89) [lower limit 0.89]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -9.1, 95% CI 2-sided [-11.26 to -6.89]

28. Secondary Outcome: Part B: Percent Change From Baseline in SCORing Atopic Dermatitis (SCORAD) at Week 16
Description: The SCORAD index is a clinical tool for assessing the severity of atopic dermatitis (AD). Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease). A negative change from baseline indicated improvement.
Time Frame: Week 16
Population: as for outcome 26
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 79 | 83
Percent Change | -16.2 (3.54) [lower limit 3.54] | -54.7 (3.39) [lower limit 3.39]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -38.4, 95% CI 2-sided [-46.65 to -30.21]

29. Secondary Outcome: Part B: Change From Baseline in Participant's Sleep Quality NRS at Week 16
Description: A sleep diary is completed by the parent/caregiver, included 2 questions assessing the caregiver's sleep, and 6 questions assessing the child's sleep based on caregiver observation. Sleep diary items, either alone or in combination serve as subjective measures of sleep quality, difficulty falling asleep, nighttime awakenings, and sleep duration. Sleep quality is measured using an 11-point NRS (0 to 10) in which 0 indicates worst possible sleep while 10 indicates best possible sleep.
Time Frame: Week 16
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 79 | 83
Score on a Scale | 0.34 (0.256) [lower limit 0.256] | 2.04 (0.251) [lower limit 0.251]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, ANCOVA — Threshold significance was at 0.05 level; LS Mean Difference = 1.70, 95% CI 2-sided [1.093 to 2.317]

30. Secondary Outcome: Part B: Change From Baseline in Participant's Skin Pain NRS at Week 16
Description: Skin pain was assessed by the parent/caregiver and measured using a 11-point scale (0 to 10) in which 0 indicated no pain while 10 indicated worst pain possible. A negative change from baseline indicated improvement.
Time Frame: Week 16
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 79 | 83
Score on a Scale | -0.62 (0.302) [lower limit 0.302] | -3.93 (0.295) [lower limit 0.295]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, ANCOVA — Threshold significance at 0.05 level; LS Mean Difference = -3.31, 95% CI 2-sided [-4.029 to -2.600]

31. Secondary Outcome: Part B: Change From Baseline in Dermatitis Family Index (DFI) at Week 16
Description: DFI is a 10-item questionnaire with items inquiring about housework, food preparation, sleep, family leisure activity, shopping, expenditure, tiredness, emotional distress, relationships, and impact of helping with treatment on the primary caregiver's life. DFI questions were scored on a four-point Likert scale ranging from 0 to 3, so that the total DFI score ranges from 0 to 30. Timeframe of reference was the past week. A higher DFI score indicated greater impairment in family Quality of life (QOL) as affected by atopic dermatitis. A negative change from baseline indicated improvement.
Time Frame: Week 16
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 79 | 83
Score on a Scale | -2.68 (0.839) [lower limit 0.839] | -10.48 (0.806) [lower limit 0.806]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, ANCOVA — Threshold significance at 0.05 level; LS Mean Difference = -7.80, 95% CI 2-sided [-9.789 to -5.814]

32. Secondary Outcome: Part B: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) at Week 16
Description: CDLQI is a validated 10 question tool to measure impact of skin disease on QOL in children by assessing how much the skin problem has affected the subjects over past week. Nine questions were scored as follows: Very much = 3, Quite a lot = 2, Only a little = 1, Not at all or unanswered = 0. Question 7 has an added possible response, which was scored as 3. CDLQI equals the sum of the score of each question (max. = 30, min. = 0). Higher the score, the greater the impact on QOL. A negative change from baseline indicated improvement.
Time Frame: Week 16
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 38 | 47
Score on a Scale | -2.5 (1.66) [lower limit 1.66] | -10.0 (1.56) [lower limit 1.56]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, ANCOVA — Threshold significance at 0.05 level; LS Mean Difference = -7.5, 95% CI 2-sided [-10.29 to -4.75]

33. Secondary Outcome: Part B: Change From Baseline in Infants' Dermatology Quality of Life Index (IDQOL) at Week 16
Description: Infants' Dermatitis Quality of Life Index (IDQOL) is used to evaluate quality of life for subjects of age less than 4 years. IDQOL questionnaires were designed for infants (below the age of 4 years) with atopic dermatitis. The IDQOL was calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score in each questionnaire, the more quality of life is impaired. A negative change from baseline indicated improvement.
Time Frame: Week 16
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 41 | 36
Score on a Scale | -1.95 (1.078) [lower limit 1.078] | -10.91 (1.159) [lower limit 1.159]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p < 0.0001, ANCOVA — Threshold significance at 0.05 level; LS Mean Difference = -8.96, 95% CI 2-sided [-11.711 to -6.202]

34. Secondary Outcome: Part B: Percentage of Topical Corticosteroid (TCS) Medication-free Days From Baseline to Week 16
Description: Percentage of TCS medication-free days was calculated as the number of days that a subject used neither TCS/TCI nor system rescue therapy divided by the study days.
Time Frame: Baseline up to Week 16
Population: The FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized).
Measure: Median (Full Range); unit: Percentage of Days
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 77 | 82
Percentage of Days | 0.04 (0.0) [0.0 to 0.9] | 0.21 (0.0) [0.0 to 1.0]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p = 0.0015, ANCOVA — Threshold significance is at 0.05 level

35. Secondary Outcome: Part B: Mean Weekly Dose of Low Potency TCS in Grams From Baseline to Week 16
Description: Mean weekly dose of TCS in grams/week for low potency TCS from baseline to Week 16 is reported.
Time Frame: Baseline up to Week 16
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: Grams per Week
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 78 | 81
Grams per Week | 13.4 (1.44) [lower limit 1.44] | 10.5 (1.39) [lower limit 1.39]
Statistical Analysis 1: Comparison: Part B: Placebo + TCS vs Part B: Dupilumab 200 mg or 300 mg Q4W + TCS; Test type: Superiority; p = 0.0997, ANCOVA — Threshold significance at 0.05 level; LS Mean Difference = -2.9, 95% CI 2-sided [-6.35 to 0.56]

36. Secondary Outcome: Part B: Mean Weekly Dose of TCS in Grams for Medium or High Potency TCS From Baseline to Week 16
Description: Mean weekly dose of TCS in grams/week for medium or high potency TCS from baseline to Week 16 is reported.
Time Frame: Baseline up to Week 16
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: Grams per Week
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 43 | 24
Grams per Week | 6.1 (1.70) [lower limit 1.70] | 3.0 (1.54) [lower limit 1.54]

37. Secondary Outcome: Part B: Mean Number of Caregiver Missed Work Days Through Week 16
Description: Mean of number of caregiver missed work days through Week 16 is reported.
Time Frame: Baseline through Week 16
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
Number analyzed (Participants) | 57 | 57
Days | 5.05 (8.975) [lower limit 8.975] | 2.49 (5.524) [lower limit 5.524]

ADVERSE EVENTS:
Time Frame: From day of first treatment up to Week 28 (end of study)
Arm/Group | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg | Part B: Placebo + TCS | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/78 | 0/83
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 1/10 | 0/10 | 4/78 | 0/83
Other Adverse Events (participants affected / at risk) | 7/10 | 7/10 | 3/10 | 2/10 | 45/78 | 29/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg (N=10) | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg (N=10) | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg (N=10) | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg (N=10) | Part B: Placebo + TCS (N=78) | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS (N=83)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 3 mg/kg (N=10) | Part A: Cohort 1 (≥2 to <6 Years Old): Dupilumab 6 mg/kg (N=10) | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 3 mg/kg (N=10) | Part A: Cohort 2 (≥6 Months to <2 Years): Dupilumab 6 mg/kg (N=10) | Part B: Placebo + TCS (N=78) | Part B: Dupilumab 200 mg or 300 mg Q4W + TCS (N=83)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 7 (8) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 7 (9) | 5 (5)
Impetigo (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 6 (7) | 3 (3)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 24 (46) | 12 (17)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 3 (3)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 5 (6) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 7 (9) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT03346434/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT03346434/SAP_001.pdf